CLINICAL TRIAL: NCT03507335
Title: Chest Strap and PPG-device Compared to Holter-device for Atrial Fibrillation Detection: 24 Hour Study
Brief Title: Atrial Fibrillation Detection: 24 Hour Study
Acronym: AFIB24h
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Tero Martikainen, Chief physician, Kuopio University Hospital
Other Study IDs: KUH507P001
Record Dates: First submitted 2017-12-20; First posted 2018-04-25 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Arrhythmia Atrial; Stroke
Keywords: Arrhythmia Atrial; heart rate monitoring; stroke; atrial fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Atrial fibrillation: Patients with atrial fibrillation during measurements
  Interventions: Device: chest strap and PPG-device for monitoring the rhythm
- Sinus: Patients with sinus rhythm during measurements
  Interventions: Device: chest strap and PPG-device for monitoring the rhythm

INTERVENTIONS:
Device: chest strap and PPG-device for monitoring the rhythm — chest strap and PPG-device for monitoring the rhythm during 24 hours for both groups (atrial fibrillation and sinus)
  Other Names: Suunto Movesense, Suunto, Vantaa, Finland; Empatica Empatica ltd, Milan, Italy

SUMMARY:
Aims Approximately 20-25% of strokes are of cardioembolic origin, atrial fibrillation (AF) being a significant cause of cardioembolic strokes. AF is often symptomless and intermittent, making its detection a clinical challenge. Currently the golden standard for diagnosis of AF is by 12-lead electrocardiogram (ECG) or any other ECG-strip.

The primary aim of the study is to assess the potential of chest strap as an ECG monitor especially in arrhythmia detection by cardiologist and algorithm. The secondary aim is to assess potential of photoplethysmography (PPG) based device for arrhythmia detection.

DETAILED DESCRIPTION:
Study design:

Study design will be a prospective case-control study at Kuopio University Hospital (KUH) in Finland. Study material will be collected in internal medicine emergency department at KUH. The study design was approved by University of Eastern Finland ethics committee (347/2018).

Study participants will receive a written information sheet about the study and will be provided with an opportunity to ask questions concerning the study. A written informed consent will be signed by the participants, including a permission to use patient's medical records.

Screening of study participants will be made in participating hospitals from admitted patients in January 2018 - May 2019. The inclusion criteria for study group patients was atrial fibrillation confirmed by a doctor-interpreted 12-lead ECG . Exclusion criteria were: body mass index (BMI) over 35; implanted pacemaker device; 12-lead ECG findings of left bundle branch block (LBBB) or right bundle branch block (RBBB); medical condition requiring immediate treatment that would be delayed by the study measurements; serious infectious disease. Control group consisted of patients with normal sinus rhythm (SR) in 12-lead ECG.

Measurement

Demographics of study patients, including age, gender, previous medical history (as reported by patient or from patient medical records), length and weight , will be recorded.

Before measurements, the patient will be asked to rest for at least 2 minutes, and lay still during the measurements. First, a 12-lead ECG will taken over a period of 10 seconds for rhythm confirmation for study grouping. In the next step, altogether 5 wet electrodes will be attached to patient to record ECG with Faros 360 Holter device (Mega Elektroniikka, Kuopio, Finland) to be used as golden standard for rhythm monitoring. Simultaneously a heart rate monitoring chest strap (Suunto Movesense, Suunto, Vantaa, Finland) will applied to chest approximately 2 cm below the lower end of sternum, according to manufacturer's instructions. PPG-device (Empatica Empatica ltd, Milan, Italy) will be connected to non-dominating wrist. A total of 24 hous recording will be made. The data from heart rate chest strap will sent via Bluetooth connection to study computer; the data from Faros Holter device was recorded to device´s internal memory card and transferred to analyzing software. The data collected was anonymized and ECG data from chest strap and Holter device was analyzed using MATLAB software.

The quality of the ECG-strip will be defined as good (no or only minor artefacts), average (artefacts but QRS complex and/or P-wave identifiable) or poor (major artefacts, no identifiable QRS complex and/or P-wave) by the cardiologist. The rhythm from the ECG-strips was divided to three categories: sinus rhythm, atrial fibrillation or other/inconclusive. The cardiologists also assessed the possibility to detect P-waves from the ECG-strips with SR (yes/no).

The study population will consisted of total 200 patients. According to the initial 12-lead ECG, total 100 patients with atrial fibrillation will be collected, and control group will consist of 100 patients with normal sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

Atrial fibrillation in 12-lead ECG and admission to hospital (n=50) Sinus rhythm in 12-lead ECG and admission to hospital (n=50)

Exclusion Criteria:

* BMI>35
* LBBB
* RBBB
* medical condition requiring immediate treatment
* serious infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study material will be collected in internal medicine emergency department of KUH
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Chest strap data quality | 24 hours
  Is chest strap ECG non-inferior or superior for the atrial fibrillation detection as compared to Holter recording. Measures for determining outcome; sensitivity and specificity for the atrial fibrillation detection.

SECONDARY OUTCOMES:
Data quality to enable arrhythmia diagnosis | 24 hours
  Is photoplethysmographic measurement non-inferior or superior for the atrial fibrillation detection as compared to Holter recording. Measures for determining outcome; sensitivity and specificity for the atrial fibrillation detection.

CONTACTS AND LOCATIONS:
Overall Officials: Tero J Martikainen, PhD, Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, East-Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Europace. 2016 Nov;18(11):1609-1678. doi: 10.1093/europace/euw295. Epub 2016 Aug 27. No abstract available. PMID 27567465
- [Background] Nemati S, Ghassemi MM, Ambai V, Isakadze N, Levantsevych O, Shah A, Clifford GD. Monitoring and detecting atrial fibrillation using wearable technology. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3394-3397. doi: 10.1109/EMBC.2016.7591456. PMID 28269032
- [Background] Thijs V. Atrial Fibrillation Detection: Fishing for An Irregular Heartbeat Before and After Stroke. Stroke. 2017 Oct;48(10):2671-2677. doi: 10.1161/STROKEAHA.117.017083. Epub 2017 Sep 15. No abstract available. PMID 28916671
- [Background] Mairesse GH, Moran P, Van Gelder IC, Elsner C, Rosenqvist M, Mant J, Banerjee A, Gorenek B, Brachmann J, Varma N, Glotz de Lima G, Kalman J, Claes N, Lobban T, Lane D, Lip GYH, Boriani G; ESC Scientific Document Group. Screening for atrial fibrillation: a European Heart Rhythm Association (EHRA) consensus document endorsed by the Heart Rhythm Society (HRS), Asia Pacific Heart Rhythm Society (APHRS), and Sociedad Latinoamericana de Estimulacion Cardiaca y Electrofisiologia (SOLAECE). Europace. 2017 Oct 1;19(10):1589-1623. doi: 10.1093/europace/eux177. No abstract available. PMID 29048522
- [Result] Freedman B, Camm J, Calkins H, Healey JS, Rosenqvist M, Wang J, Albert CM, Anderson CS, Antoniou S, Benjamin EJ, Boriani G, Brachmann J, Brandes A, Chao TF, Conen D, Engdahl J, Fauchier L, Fitzmaurice DA, Friberg L, Gersh BJ, Gladstone DJ, Glotzer TV, Gwynne K, Hankey GJ, Harbison J, Hillis GS, Hills MT, Kamel H, Kirchhof P, Kowey PR, Krieger D, Lee VWY, Levin LA, Lip GYH, Lobban T, Lowres N, Mairesse GH, Martinez C, Neubeck L, Orchard J, Piccini JP, Poppe K, Potpara TS, Puererfellner H, Rienstra M, Sandhu RK, Schnabel RB, Siu CW, Steinhubl S, Svendsen JH, Svennberg E, Themistoclakis S, Tieleman RG, Turakhia MP, Tveit A, Uittenbogaart SB, Van Gelder IC, Verma A, Wachter R, Yan BP; AF-Screen Collaborators. Screening for Atrial Fibrillation: A Report of the AF-SCREEN International Collaboration. Circulation. 2017 May 9;135(19):1851-1867. doi: 10.1161/CIRCULATIONAHA.116.026693. PMID 28483832
- [Derived] Santala OE, Lipponen JA, Jantti H, Rissanen TT, Tarvainen MP, Laitinen TP, Laitinen TM, Castren M, Valiaho ES, Rantula OA, Naukkarinen NS, Hartikainen JEK, Halonen J, Martikainen TJ. Continuous mHealth Patch Monitoring for the Algorithm-Based Detection of Atrial Fibrillation: Feasibility and Diagnostic Accuracy Study. JMIR Cardio. 2022 Jun 21;6(1):e31230. doi: 10.2196/31230. PMID 35727618
- [Derived] Santala OE, Halonen J, Martikainen S, Jantti H, Rissanen TT, Tarvainen MP, Laitinen TP, Laitinen TM, Valiaho ES, Hartikainen JEK, Martikainen TJ, Lipponen JA. Automatic Mobile Health Arrhythmia Monitoring for the Detection of Atrial Fibrillation: Prospective Feasibility, Accuracy, and User Experience Study. JMIR Mhealth Uhealth. 2021 Oct 22;9(10):e29933. doi: 10.2196/29933. PMID 34677135